CLINICAL TRIAL: NCT05096923
Title: UNC Childhood, Adolescent, and Young Adult Cancer Cohort
Acronym: UNC-CAYACC
Status: Recruiting | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Hyundai Hope On Wheels (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC 2116
Record Dates: First submitted 2021-10-14; First posted 2021-10-27 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Pediatric Cancer; Cancer; Cancer Metastatic; Survivorship
Keywords: Adolescent and young adult; AYA
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples With DNA — Up to 22.5 milliliters of peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UNC-CAYACC: Children, adolescents, and young adults diagnosed with cancer before the age of 40 enrolled at any point during the diagnosis-treatment-survivorship continuum.

SUMMARY:
Purpose: This study aims to create a registry of childhood, adolescent, and young adult patients with cancer (<40 years-old at cancer diagnosis), entitled the 'UNC Childhood, Adolescent, and Young Adult Cancer Cohort' (UNC-CAYACC). This resource will serve to support cancer outcomes research among pediatric and young adult cancer patients with a primary focus on enrolling patients treated as adolescents or young adults (AYAs, 15-39 years).

Procedures: As appropriate for age, participants will complete physical and cognitive functional assessments; questionnaires to assess health-related quality of life and other patient-reported outcomes; will undergo body composition and anthropometric measurements; and will be asked to provide biospecimens for biobanking. Assessments will be collected (as possible) at diagnosis, during active treatment, following treatment completion, and annually in survivorship to assess outcomes throughout the treatment and survivorship trajectory. Sociodemographic and clinical information such as cancer treatment modalities and cumulative doses will be collected by medical record abstraction. Participants will be eligible to enroll at any time from diagnosis through survivorship. This registry will provide data to better understand the manifestations of accelerated aging and key contributing factors among children, adolescents, and young adults with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient ages 0-39 years at the time of cancer diagnosis (ages 1-39 years at enrollment) who are at any point in treatment and survivorship trajectory
* English or Spanish speaking

Exclusion Criteria:

* Unwilling to sign informed consent
* Speak a language other than English or Spanish.

Ages: 1 Year to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Child, adolescent, and young adult (0-39 years-old at diagnosis, 1-39 years at enrollment) patients with cancer who will undergo or have undergone treatment or receive follow up care at the NC Children's Hospital, the NC Cancer Hospital, or one of the UNC Health affiliated clinical sites.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-12-17 (Actual); Primary Completion 2031-01-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Registry development | Five years
  Creation of a registry of pediatric and young adult patients with cancer treated within the University of North Carolina Health System
Functional assessments | Five years
  Assess feasibility for completing repeated physical and cognitive functional assessments among young cancer survivors. These assessments include measures of physical and general frailty.

SECONDARY OUTCOMES:
Collection of sociodemographic, cancer, and treatment variables | Five years
  Assess feasibility for collection of sociodemographic (including social determinants of health), cancer (e.g., site and stage), and treatment (e.g., modalities and cumulative doses) variables using patient questionnaires and medical record abstraction.
Collection of patient-reported outcome measures | Five years
  Assess feasibility for the repeated collection of patient-reported measures of health-related quality of life, health behaviors, and functional status.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Smitherman, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified aggregate data will be available upon request. De-identified or coded individual data from the registry may be made available upon request following completion of necessary data use agreements and with Institutional Review Board (IRB) approval.
Access Criteria: Data use inquiries should be directed to Andrew Smitherman, MD at andrew_smitherman@med.unc.edu. Requests will be reviewed and final decisions on release of data made by the UNC-CAYACC Governance and Data Sharing Committee.